CLINICAL TRIAL: NCT04281147
Title: Real World Evaluation of Access-driven Canadian Treatment Sequences in Progressive Prostate Cancer
Brief Title: Study to Gather Information About the Use of Healthcare Services and the Way the Disease is Cared for in Canadian Patients With Prostate Gland Cancer Which Spread Throughout the Body
Acronym: REACTIVATE
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20949
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer
Keywords: Metastatic castrate resistant prostate cancer mCRPC
MeSH Terms: conditions — Prostatic Neoplasms | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No Ra-223 received: Patients did not receive Ra-223
- Early Ra-223 (2nd line): Patients received Ra-223 in 2nd line
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223)
- Late Ra-223 (3rd or later lines): Patients received Ra-223 in 3rd or later lines
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223)

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY88-8223) — Follow clinical administration
  Groups: Early Ra-223 (2nd line); Late Ra-223 (3rd or later lines)

SUMMARY:
Study to gather information about the optimal placement of Ra-223 in the order of different treatments in terms of the effect on patients and in terms of the use of healthcare services for the treatment of Canadian patients with prostate gland cancer which spread to other parts of the body. In order to collect this information real world data from prostate gland cancer patients from four Canadian administrative databases will be analyzed.

Data collected from patients treated with their 2nd line of life-prolonging therapy for Non-Metastatic Castration Resistant Prostate Cancer (mCRPC) initiated from 01 Jan 2012 to 31 Dec 2017. For patients included in the study, all available data from the beginning for their record until death, lost to follow-up or database cut-off will be included. The index date is the date of initiation of the 2nd line life-prolonging therapy for mCRPC.

ELIGIBILITY:
Inclusion Criteria:

* Use of at least 2 lines of life-prolonging mCRPC therapy
* The 2nd line of life-prolonging therapy was initiated between 01-Jan-2012 to 31-Dec-2017

Exclusion Criteria:

- No formal exclusion criteria will be applied in order to capture real world use of Ra-223

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men with mCRPC and at least 2 lines of life-prolonging therapy initiated between 01 Jan 2012 to 31 Dec 2017. No formal exclusion criteria will be applied in order to capture real world use of Ra-223.
Sampling Method: Non-Probability Sample
Enrollment: 4301 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Overall survival | Retrospective analysis from 01-Jan-2012 to 31-Dec-2017
  The length of time from the date of initiation of 2nd line life-prolonging therapy to death due to any cause

SECONDARY OUTCOMES:
Event-free survival (EFS) | Retrospective analysis from 01-Jan-2012 to 31-Dec-2017
  The length of time from the start of 2nd line life-prolonging therapy to the earliest occurrence of one of the following:
  * A change in life-prolonging treatment
  * Death from any cause
Time to External Beam Radiation Therapy (EBRT) | Retrospective analysis from 01-Jan-2012 to 31-Dec-2017
  From the start of the 1st life-prolonging therapy (index date) until the first use of EBRT
Total incidence of EBRT | Retrospective analysis from 01-Jan-2012 to 31-Dec-2017
  Total number of EBRT treatments received over the course of the patient's journey starting from the initiation of 2nd line life-prolonging therapy (index date) until death.
Time to first hospitalization | Retrospective analysis from 01-Jan-2012 to 31-Dec-2017
  Measured from the start of the 2nd line life-prolonging therapy (index date) until the first overnight hospital stay.
Number of overnight hospital stays | Retrospective analysis from 01-Jan-2012 to 31-Dec-2017
  Measured from the initiation of 2nd line life-prolonging therapy (index date) until death
Average length of hospital stays (number of days) | Retrospective analysis from 01-Jan-2012 to 31-Dec-2017
  Measured from the initiation of 2nd line life -prolonging therapy (index date) until death
Time to first Emergency Room (ER) visit | Retrospective analysis from 01-Jan-2012 to 31-Dec-2017
  Measured from the start of 2nd line life-prolonging therapy (index date) until the first ER visit.
Number of visits to the ER | Retrospective analysis from 01-Jan-2012 to 31-Dec-2017
  Measured from the initiation of 2nd line life-prolonging therapy (index date) until death

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple Locations, Multiple Locations, Canada

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.